CLINICAL TRIAL: NCT07022730
Title: The Novel Use of Prophylactic Noradrenaline Infusion and Its Impact on Post-induction Hypotension in Patients With Surgical Sepsis, a Double Blind Randomized Controlled Trial
Brief Title: Prophylactic Noradrenaline Infusion and Its Impact on Post-induction Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: noradrenaline and PIH
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Post Induction Hypotension; Sepsis
Keywords: Hypotension; noradrenaline; sepsis
MeSH Terms: conditions — Sepsis; Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noradrenaline (Active Comparator): Noradrenaline will be infused at a fixed rate of 0.2 mic/kg/min at 5 minutes before induction
  Interventions: Drug: Noradrenaline 0.2 mcg/kg/min at 5 minutes before induction
- Control (No Intervention): Patients will receive normal saline

INTERVENTIONS:
Drug: Noradrenaline 0.2 mcg/kg/min at 5 minutes before induction — noradrenaline will be given at a rate of 0.2 mcg/kg/min that will start 5 minutes before induction
  Arms: Noradrenaline

SUMMARY:
researchers aim to evaluate the influence of prophylactic noradrenaline infusion on post-induction hypotension

DETAILED DESCRIPTION:
If post-induction hypotension is not addressed promptly, it can lead to severe complications such as reduced blood flow, acute kidney damage, and myocardial ischemia. As a result, early detection and proactive intervention are crucial. Researchers of the current study decided to investigate impact of noradrenaline administered as a prophylaxis on post induction hypotension

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with sepsis undergoing source control surgery.

Exclusion Criteria:

* Patient refusal
* Patient with cardiac pathology ( ischemic heart disease or heart failure)
* Preoperative hemodynamic instability (defined as MAP < 65 mmHg)
* Rapid sequence induction

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-06-22 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Incidence of post induction hypotension in both groups | Within the first 10 minutes of induction.
  Hypotension will be considered if MAP< 65 mmHg

SECONDARY OUTCOMES:
Incidence of acute kidney injury | 7 days post operative
  defined as the highest postoperative value > 1.5-fold or 0.3 mg/dL greater than the preoperative value
Incidence of myocardial infarction | 7 days postoperative
  defined as a peak troponin T value exceeding 15 times the normal upper limit, along with new pathological Q waves, ST elevation or depression, and hyperacute T wave on ECG and symptoms suggestive of myocardial infarction
Incidence of stroke | 7 days postoperative
  clinical or image finding of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to privacy concerns, regulatory restrictions, and informed consent limitations.

REFERENCES:
- [Background] Goertz AW, Lindner KH, Seefelder C, Schirmer U, Beyer M, Georgieff M. Effect of phenylephrine bolus administration on global left ventricular function in patients with coronary artery disease and patients with valvular aortic stenosis. Anesthesiology. 1993 May;78(5):834-41. doi: 10.1097/00000542-199305000-00005. PMID 8489054
- [Background] Czajka S, Putowski Z, Krzych LJ. Post-induction hypotension and intraoperative hypotension as potential separate risk factors for the adverse outcome: a cohort study. J Anesth. 2023 Jun;37(3):442-450. doi: 10.1007/s00540-023-03191-7. Epub 2023 Apr 21. PMID 37083989
- [Background] Tangkulpanich P, Angkoontassaneeyarat C, Trainarongsakul T, Jenpanitpong C. Factors Associated with Postintubation Hypotension Among Patients with Suspected Sepsis in Emergency Department. Open Access Emerg Med. 2023 Nov 14;15:427-436. doi: 10.2147/OAEM.S426822. eCollection 2023. PMID 38022743